CLINICAL TRIAL: NCT06330922
Title: Muscle-tendon Pathology, Metabolic Dysregulation and Chronic Inflammation in Adolescents and Young Adults With Moderate to Severe Spastic Cerebral Palsy
Brief Title: Muscle-tendon Pathology and Metabolic Dysregulation in CP
Status: Recruiting | Type: Observational
Sponsor: University of Graz (Other)
Collaborators: Medical University of Graz (Other); Karolinska Institutet (Other)
Responsible Party: Sponsor
Other Study IDs: 10.55776/V992
Record Dates: First submitted 2024-03-11; First posted 2024-03-26 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Cerebral Palsy, Spastic
Keywords: Cerebral Palsy; Spasticity; Cardiorespiratory Fitness; Frame Running; Muscle
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Where applicable, serum and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: healthy individuals (cross-sectional study): Typically developed adolescents and young adults will be recruited and measured once within the cross-sectional study.
- Group 2: mildly affected individuals with cerebral palsy (cross-sectional study): Mildly affected adolescents and young adults will be recruited and measured once within the cross-sectional study.
- Group 3: moderately and severely affected individuals with cerebral palsy (cross-sectional study): The results of the baseline assessment (T0) of the adolescents and young adults with moderate to severe cerebral palsy will be compared with group 1 and group 2.
  After the baseline assessment (T0) also used for the group comparison (see description above), group 3 enters a 12-week control period following daily routines. After the 12 weeks, the individuals will be assessed (T1) and will then start with the 12-week cardiorespiratory fitness training. The final assessment (T2) will terminate study participation of group 3.
  Interventions: Other: Cardiorespiratory fitness training

INTERVENTIONS:
Other: Cardiorespiratory fitness training — Cardiorespiratory fitness training will be performed two times a week for one hour in small groups (4-5 people). The training will be conducted outdoors at track and field facilities with at least two coaches.
  Other Names: Frame Running
  Groups: Group 3: moderately and severely affected individuals with cerebral palsy (cross-sectional study)

SUMMARY:
The main aim of this project is to gain knowledge about the muscle-tendon pathology of moderately to severely affected young people with cerebral palsy and their risk for cardiometabolic diseases and chronic inflammation. Furthermore, it will be investigated whether there are associations between the existing pathophysiology as well as inactivity and muscle function, cardiometabolic risk factors and inflammation. Moreover, the potential of the target group for adaptation of its muscular, cardiorespiratory, and endocrine system will be investigated.

The study parameters will be determined in adolescents and young adults aged 14 to 30 years with moderate to severe spastic cerebral palsy and compared with those of their less severely affected and healthy peers (cross-sectional study). In addition, the more affected individuals will participate in a 12-week training intervention (longitudinal study) performed with special tricycles (i.e., Frame Runners).

To measure the study parameters, ultrasound, strength tests, near-infrared spectroscopy, blood analyses, and spiroergometry will be used. The fitness training will be performed two times a week for 12 weeks with the Frame Runners.

DETAILED DESCRIPTION:
Background: Spastic cerebral palsy (CP) is a neuro-developmental disorder in children. Although the initial brain injury is not progressive, muscle pathology, a leading sign in affected individuals, is an on-going process. Individuals with CP are less physically active compared to their typically developing (TD) peers and severely affected individuals are most sedentary. Therefore, increased muscle wasting, decreased muscle function and cardiorespiratory fitness, metabolic dysregulation, and chronic low-grade inflammation might exist in the latter group. However, information is scarce and the role of muscle-tendon pathology and physical inactivity remains to be elucidated. Finally, it is unknown whether their tissues and organs may still adapt to health-inducing stimuli.

Objectives: The main project aims are 1) to enhance our understanding of spastic muscle-tendon pathology, risk of cardiometabolic disease, and chronic inflammation likely present in young people with more severe spastic CP, and 2) to uncover the relationship of muscle-tendon alterations and physical inactivity on muscle function and metabolism as well as cardiometabolic risk factors and systemic inflammation. Moreover, the potential for adaptation of their muscular, cardiorespiratory, and endocrine system will be investigated.

Methods: A cross-sectional study will be performed to compare severely impaired adolescents and young adults with spastic CP, their mildly affected CP and TD peers. The former group will further participate in a 12-week cardiorespiratory fitness training with Frame Runners. Muscle properties will be examined using ultrasound and shear wave elastography, and muscle function and metabolism with dynamometry and near infrared spectroscopy. Blood samples will be analyzed assessing metabolic parameters, and pro-inflammatory cytokines. Cardiorespiratory fitness will be investigated using the 6-Minute Frame Running Test and gas exchange analysis. Physical activity will be evaluated with accelerometers and activity diaries. Mental well-being and quality of life will be assessed by use of the CPCHILD™ questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* spastic cerebral palsy
* mildly, moderately or severly affected (Gross Motor Function Classification System level I-IV)
* age range 14 - 30 years
* ability to accept and follow verbal instructions
* strong communication skills
* sufficient vision (visual function that enables safe movement with reference to people and obstacles)
* less than 15 hours of experience with the Frame Runners; healthy peers in the same age range

Exclusion Criteria:

* other forms of cerebral palsy
* orthopaedic surgery in the last 12 months
* Botulinum toxin application in the last 6 months

Ages: 14 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The patient selection is based on the inclusion and exclusion criteria from the patient pool of the local clinic for Orthopaedics and Traumatology. In addition, other interested persons/families will be informed about the study via other clinics, (pediatric orthopedic) elective medical practices, rehabilitation centers and physiotherapy facilities within the city and the surrounding area.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Muscle fascicle length and muscle thickness | Group 1 & 2: baseline (T0); Group 3: baseline (T0), pre-measurement (T1, 13 weeks), post-measurement (T2, 27 weeks)
  cm
Muscle fascicle pennation angle | Group 1 & 2: baseline (T0); Group 3: baseline (T0), pre-measurement (T1, 13 weeks), post-measurement (T2, 27 weeks)
  degrees
Passive muscle stiffness | Group 1 & 2: baseline (T0); Group 3: baseline (T0), pre-measurement (T1, 13 weeks), post-measurement (T2, 27 weeks)
  kilopascal (kPa)
Isometric muscle strength | Group 1 & 2: baseline (T0); Group 3: baseline (T0), pre-measurement (T1, 13 weeks), post-measurement (T2, 27 weeks)
  kg
Muscle tissue oxygenation | Group 1 & 2: baseline (T0); Group 3: baseline (T0), pre-measurement (T1, 13 weeks), post-measurement (T2, 27 weeks)
  Tissue saturation index (TSI)
Exosome size | Group 1 & 2: baseline (T0); Group 3: baseline (T0), pre-measurement (T1, 13 weeks), post-measurement (T2, 27 weeks)
  nanometers (nm)
Exosome content | Group 1 & 2: baseline (T0); Group 3: baseline (T0), pre-measurement (T1, 13 weeks), post-measurement (T2, 27 weeks)
  number/ml
Micro ribonucleic acid (RNA) cargo | Group 1 & 2: baseline (T0); Group 3: baseline (T0), pre-measurement (T1, 13 weeks), post-measurement (T2, 27 weeks)
  expression level

SECONDARY OUTCOMES:
Metabolic parameters | Group 1 & 2: baseline (T0); Group 3: baseline (T0), pre-measurement (T1, 13 weeks), post-measurement (T2, 27 weeks)
  Glucose, C-peptide, free fatty acids, cholesterol, triglycerides, high-density lipoprotein, low-density lipoprotein in mmol/l
Pro-inflammatory cytokines | Group 1 & 2: baseline (T0); Group 3: baseline (T0), pre-measurement (T1, 13 weeks), post-measurement (T2, 27 weeks)
  e.g., Interleukin 6, tumor necrosis factor alpha in pg/ml
Resting, mean, and peak heart rate | Group 1 & 2: baseline (T0); Group 3: baseline (T0), pre-measurement (T1, 13 weeks), measurement after 6 weeks of training (T1_6weeks, 20 weeks), post-measurement (T2, 27 weeks)
  beats/min
Resting blood pressure | Group 1 & 2: baseline (T0); Group 3: baseline (T0), pre-measurement (T1, 13 weeks), post-measurement (T2, 27 weeks)
  mmHg
Distance covered | Group 1 & 2: baseline (T0); Group 3: baseline (T0), pre-measurement (T1, 13 weeks), measurement after 6 weeks of training (T1_6weeks, 20 weeks), post-measurement (T2, 27 weeks)
  m
Peak oxygen uptake (VO2peak), Peak ventilation (VEpeak) | Group 1 & 2: baseline (T0); Group 3: baseline (T0), pre-measurement (T1, 13 weeks), measurement after 6 weeks of training (T1_6weeks, 20 weeks), post-measurement (T2, 27 weeks)
  l/min
Peak respiratory frequency | Group 1 & 2: baseline (T0); Group 3: baseline (T0), pre-measurement (T1, 13 weeks), measurement after 6 weeks of training (T1_6weeks, 20 weeks), post-measurement (T2, 27 weeks)
  breaths/min
Respiratory exchange ratio | Group 1 & 2: baseline (T0); Group 3: baseline (T0), pre-measurement (T1, 13 weeks), measurement after 6 weeks of training (T1_6weeks, 20 weeks), post-measurement (T2, 27 weeks)
  peak carbon dioxide production (VCO2peak)/VO2peak
VEpeak/VO2peak | Group 1 & 2: baseline (T0); Group 3: baseline (T0), pre-measurement (T1, 13 weeks), measurement after 6 weeks of training (T1_6weeks, 20 weeks), post-measurement (T2, 27 weeks)
  ratio
VEpeak/VCO2peak | Group 1 & 2: baseline (T0); Group 3: baseline (T0), pre-measurement (T1, 13 weeks), measurement after 6 weeks of training (T1_6weeks, 20 weeks), post-measurement (T2, 27 weeks)
  ratio
Perceived exertion | Group 1 & 2: baseline (T0); Group 3: baseline (T0), pre-measurement (T1, 13 weeks), measurement after 6 weeks of training (T1_6weeks, 20 weeks), post-measurement (T2, 27 weeks)
  6-20 Borg Scale
Well-being and quality of life | Group 1 & 2: baseline (T0); Group 3: baseline (T0), pre-measurement (T1, 13 weeks), post-measurement (T2, 27 weeks)
  Caregiver Priorities and Child Health Index of Life with Disabilities (CPCHILD™) questionnaire
Total physical activity, time spent in different intensities | Group 1 & 2: within 1 week between familiarisation and baseline (T0); Group 3: within 1 week after baseline (T0), within 1 week after post-measurement (T2, 28 weeks)
  min
Passive range of motion (sagittal plane) of hip, knees, ankles | Group 1 & 2: baseline (T0); Group 3: baseline (T0), pre-measurement (T1, 13 weeks), post-measurement (T2, 27 weeks)
  degrees
Step count | Group 1 & 2: within 1 week between familiarisation and baseline (T0); Group 3: within 1 week after baseline (T0), within 1 week after post-measurement (T2, 28 weeks)
  number

OTHER OUTCOMES:
Body height | Group 1 & 2: baseline (T0); Group 3: baseline (T0), pre-measurement (T1, 13 weeks), post-measurement (T2, 27 weeks)
  cm
Body weight | Group 1 & 2: baseline (T0); Group 3: baseline (T0), pre-measurement (T1, 13 weeks), post-measurement (T2, 27 weeks)
  kg
Body mass index (BMI) | Group 1 & 2: baseline (T0); Group 3: baseline (T0), pre-measurement (T1, 13 weeks), post-measurement (T2, 27 weeks)
  Body height and weight will be combined to calculate the BMI in kg/m^2
Modified Ashworth Scale Score of the Plantar flexors | Group 2: baseline (T0); Group 3: baseline (T0), pre-measurement (T1, 13 weeks), post-measurement (T2, 27 weeks)
  number

CONTACTS AND LOCATIONS:
Overall Officials: Annika Kruse, Dr., Principal Investigator — Institute of Human Movement Science, Sport and Health, University of Graz
Locations (1):
- Institute of Human Movement Science, Sport and Health, University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Yes
Open access to research data on which the research publications are based will be provided following the Criteria for Open Research Data presented by the Austrian Science fund (FWF). If data can be shared (i.e., anonymisation can be ensured), it will be deposited under the Creative Commons (CC BY) licence.
Time Frame: Research data on which future papers are based will be made available shortly after publication.
Access Criteria: Individual participant data (IPD) will be provided under the CC BY licence.

REFERENCES:
- [Background] Bell KJ, Ounpuu S, DeLuca PA, Romness MJ. Natural progression of gait in children with cerebral palsy. J Pediatr Orthop. 2002 Sep-Oct;22(5):677-82. PMID 12198474
- [Background] Graham HK, Rosenbaum P, Paneth N, Dan B, Lin JP, Damiano DL, Becher JG, Gaebler-Spira D, Colver A, Reddihough DS, Crompton KE, Lieber RL. Cerebral palsy. Nat Rev Dis Primers. 2016 Jan 7;2:15082. doi: 10.1038/nrdp.2015.82. PMID 27188686
- [Background] Narayanan UG, Fehlings D, Weir S, Knights S, Kiran S, Campbell K. Initial development and validation of the Caregiver Priorities and Child Health Index of Life with Disabilities (CPCHILD). Dev Med Child Neurol. 2006 Oct;48(10):804-12. doi: 10.1017/S0012162206001745. PMID 16978459
- [Background] Nooijen CF, Slaman J, Stam HJ, Roebroeck ME, Berg-Emons RJ; Learn2Move Research Group. Inactive and sedentary lifestyles amongst ambulatory adolescents and young adults with cerebral palsy. J Neuroeng Rehabil. 2014 Apr 3;11:49. doi: 10.1186/1743-0003-11-49. PMID 24708559
- [Background] Verschuren O, Peterson MD, Balemans AC, Hurvitz EA. Exercise and physical activity recommendations for people with cerebral palsy. Dev Med Child Neurol. 2016 Aug;58(8):798-808. doi: 10.1111/dmcn.13053. Epub 2016 Feb 7. PMID 26853808
- [Background] Howard JJ, Herzog W. Skeletal Muscle in Cerebral Palsy: From Belly to Myofibril. Front Neurol. 2021 Feb 18;12:620852. doi: 10.3389/fneur.2021.620852. eCollection 2021. PMID 33679586